CLINICAL TRIAL: NCT06074861
Title: The Effect of a Fast-mimicking Diet on Periodontal Clinical and Systemic Response to Non-surgical Treatment of Stage III-IV Periodontitis: a Multi-centre Randomised Controlled Trial With Internal Pilot
Brief Title: Fasting-mimicking Diet and Periodontitis (FMD)
Acronym: FMD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Collaborators: Universidad Complutense de Madrid (Other); University of Santiago de Compostela (Other); Universidad de Granada (Other); Universidad de Murcia (Other); King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PER-ECL-2022-02
Record Dates: First submitted 2023-09-27; First posted 2023-10-10 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Periodontal Disease, AVDC Stage 3; Periodontal Disease, AVDC Stage 4; Periodontitis
MeSH Terms: conditions — Periodontal Diseases; Periodontitis

STUDY DESIGN:
Intervention Model Description: There will be a Test group and a Control group
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test group (Active Comparator): Patients will receive the non-surgical periodontal therapy plus three cycles of fasting-mimicking diet.
  Interventions: Procedure: Fasting-mimicking diet + non-surgical periodontal therapy
- Control group (No Intervention): Patients will receive the non-surgical periodontal therapy and will continue with their normal (and ad libitum) diet.

INTERVENTIONS:
Procedure: Fasting-mimicking diet + non-surgical periodontal therapy — Test group will receive a full-mouth non-surgical periodontal therapy (also named professional mechanical plaque removal-PMPR) and, in the same day (starting at morning), a fasting-mimicking diet (FMD) will be started (for a cycle of 5 days). Other two cycles of FMD will be followed at 45- and 85- days after treatment, respectively.
  Arms: Test group

SUMMARY:
Periodontitis (gum disease) leads to the formation of gum pockets. Its treatment involves deep cleaning of the teeth, to remove soft and hard tooth deposits under the gum line. Although in the long term this leads to improvement of the gum conditions and reduced inflammation, in the hours and days post-treatment, inflammation may increase, sometimes also associated with a high temperature. A method to reduce this response has not been found yet.

The goal of this multi-centre randomized controlled trial is to to test if a diet which acts to mimic periodic fasting can influence responses in the mouth and throughout the body after treatment of gum disease in patients with advanced gum disease but general health conditions. Five Spanish centres (Universidad Complutense de Madrid, Universidad Internacional de Catalunya, Universidad de Murcia, Universidad de Santiago de Compostela, Universidad de Granada) will perform the clinical part of the study, whereas the King's College of London (Guy's Hospital) will provide the analyses and processing of the data. Researchers will include 28 patients in total.

The main question it aims to answer is:

- Is a mimic periodic fasting (together with the classical gum treatment) effective at reducing the local and systemic inflammation provoked by the gum disease (and by the same treatment) in the short- and medium term?

Although all participants will receive the necessary gum treatment (deep cleaning), researchers will randomly assign them to one of two groups.

The test group will follow three cycles (the same day of the treatment, and 45- and 85 days after treatment) of 5 days each of a fasting-mimicking diet (FMD). The FMD program is a plant-based diet program designed to attain fasting-like effects while providing both macro- and micronutrients to minimize the burden of fasting and adverse effects. The FMD consists of 100% ingredients that are generally regarded as safe (GRAS) and comprises proprietary vegetable-based soups, energy bars, energy drinks, cracker snacks, olives, herbal teas, and supplements. All items to be consumed per day are individually boxed.

In contrast, the control group will continue with their current diet. All patients will complete dietary diaries to estimate calorie intake during this time period.

Researchers will collect blood, stool, plaque and gingival crevicular fluid samples from each patient at different time points.

Besides, they will call the patients one or two times during each FMD cycle to check that everything is proceeding properly and to solve any problems or concerns they may have. In addition, a trained registered dietitian will be available during the whole study period in case participants need some support or have doubts and/or questions.

If participants miss multiple visits (e.g. 2/3) will be considered as a drop-out and, if they develop a serious medical condition, they might be excluded from the study. However, independently from the participation into this study, each patient will have their gum disease regularly treated.

People with periodontal disease usually have a bad dietary-habits. This investigation with its holistic approach might lead people to modify their unbalanced diet due to the possible related local and systemic benefits. In addition, cycles of 5 days might consistently raise the adherence and willingness to follow such a fasting regime.

DETAILED DESCRIPTION:
Introduction

Periodontitis is a microbially-driven inflammatory disease of the periodontium. It has been shown that the periodontitis-associated inflammation is not limited to the periodontium, but may have far-reaching consequences in the rest of the body, and that this may be partly mediated by systemic spread of oral microorganisms. Steps 1 and 2 of periodontal therapy is also associated with a short-term acute phase inflammatory response, characterised by elevation of circulating acute-phase inflammatory markers, which in turn is followed, if successful, by a longer-term reduction in these molecules. In the intermediate to longer term this is accompanied by changes in other markers of peripheral vascular health alongside improvements in metabolic control lasting at least 12 months. Periodontitis is known to have a bidirectional relationship with metabolic disruption and dysregulation. A very recent work corroborated that periodontitis is associated with systemic inflammation as measured by serum C-reactive protein (CRP) levels. Furthermore, it has been reported that intensive non-surgical periodontitis treatment (steps 1 and 2) led to a progressive reduction of CRP after 90 days with a moderate increase at 180 days. It is thought that improvements in metabolic control may also improve periodontal outcomes, yet the exact mechanisms for this are not fully clear. Several human and experimental investigations have also been published concerning the possible effects of nutrition on management of periodontitis. A study on monkeys found that long-term dietary caloric restriction (diet enriched with vitamins and minerals) dampens clinical inflammation and reduces the degree of periodontal breakdown secondary to acute microbial challenge. However, in another experimental study on monkeys, long-term hypocaloric diet (30% less of daily calories intake plus vitamins and minerals) appeared to differentially reduce the production of local inflammatory mediators and the risk for inflammatory periodontal disease among males but not females. In addition, a recent systematic review on animal models concluded that macronutrients that have an effect on oxidative stress or immune system (i.e., n-3 fatty acid) seem to be important for the prevention or treatment of periodontitis. In terms of human research, a Korean group, after a four-week weight control intervention in periodontally healthy obese people, observed a reduction of matrix metalloproteinase (MMP)-8, MMP-9, and interleukin-1β (IL-1β) in gingival crevicular fluid (GCF). A German team reported that a diet consisting of low carbohydrate intake, richness in Omega 3-fatty acids and fibre, higher vitamin C and D values, reduction of animal proteins, and focused intake of nitrate-containing plants might lead to a significant reduction in periodontal and gingival inflammation, even though serological inflammatory parameters and the subgingival microbiome seem to be unaffected. More recently, a study found that there was no overall association between Western dietary patterns (characterized by a higher intake of processed meat, red meat, butter, high-fat dairy products, eggs and refined grains) or prudent dietary patterns (characterized by a higher intake of vegetables, fruit, legumes, whole grains, fish and poultry) and periodontitis; however when solely obese individuals were considered, a Western diet was related to a higher risk of periodontitis. Another very recent investigation, based on use of a dietary inflammatory index, showed that consuming a pro-inflammatory diet was associated with moderate-severe periodontitis in the U.S. general adult population. A novel mode of fasting has been introduced in order to increase patient compliance, due to the fact that people are usually not able to follow a strict diet for a long period. In particular, the fasting mimicking diet (FMD), consisting of 30-50% of the normal caloric intake for 4-7 consecutive days followed by a refeeding ad libitum period once a month, showed very promising beneficious effects in terms of reduction of risk factors for aging, diabetes, autoimmunity, cardiovascular disease, neurodegeneration and cancer. Overall, there is still uncertainty about a potential role of periodic fasting on periodontal clinical and inflammatory parameters. To our knowledge, no studies have investigated the potential effect of FMD on systemic and periodontal response after periodontitis treatment.

Objectives

The main aim of this study is to test if a fasting mimicking diet can influence the systemic and periodontal response following non-surgical periodontal therapy. The null hypothesis is that a fasting mimicking diet does not modify the local and systemic inflammatory post-treatment response.

Study Design

This is a double-blind (outcome-assessor and statistician), multi-centre, randomized clinical study with parallel groups and a 1:1 allocation ration, with internal pilot. All recruited patients will receive the same protocol for periodontal therapy (steps 1 & 2). One group (test) will be submitted to three cycles of FMD. The FMD program is a plant-based diet program designed to attain fasting-like effects while providing both macro- and micronutrients to minimize the burden of fasting and adverse effects. The FMD consists of 100% ingredients that are generally regarded as safe (GRAS) and comprises proprietary vegetable-based soups, energy bars, energy drinks, cracker snacks, olives, herbal teas, and supplements. All items to be consumed per day are individually boxed to allow the subjects to choose when to eat while avoiding accidentally consuming components of the following day. The FMD consists of a 5-days regimen that provides approximately 1.100 kilocalories for the first day; approximately 750 kilocalories per day for the second to the fifth day. On the contrary, the other group (control) will continue with their normal diet.

Subject selection

This is a multi-centre study. Participants will be screened by International University of Catalunya (UIC), Complutense University of Madrid (UCM), University of Santiago de Compostela, University of Murcia and University of Granada clinical staff/students among periodontitis patients attending the respective hospitals. The investigators expect 28 eligible participants available per year and assume that 70% of them will agree to take part in the trial after expressing initial interest.

Study procedures

Subject recruitment

International University of Catalunya's, Complutense University, Santiago de Compostela and Granada Universities' patients, will be individually approached for recruitment on campus and within the Dental faculty. After expressing an initial interest, potential participants will be provided with an information sheet and the opportunity to ask questions to members of the study team via email or telephone. If they then express a desire to participate, they will be invited to a screening visit. Each individual will be given at least 24 hours and up to a week to decide if they would wish to take part. Individuals will be reimbursed for their time with a payment at completion of the study.

Screening Procedures

At the screening visit, consent will be sought by the trained applicant or study dentist, which will be recorded through a written participant consent form detailing the complete trial procedure and an agreement checklist for each data collection method. Once consent is given, each enrolled participant will be recorded on a Participant Log form. Initial screening will be to ensure that each individual conforms to the outlined inclusion and exclusion criteria. This will be assessed by taking an oral history and will be recorded on a hardcopy Screening Log form. Participants will need to undergo a periodontal examination from the study dentist to ensure suitability.

Randomisation Procedures and allocation concealment

Initial central randomization will be done using the "Sealed Envelope" method by personnel not directly involved in the study, at Guy's Hospital. For important influencing factors ('centre') stratified randomisation will be carried out as recommended. No stratification by age will be carried out, because for small sample sizes, stratification should be limited to one or very few factors and because the influence of age is limited by the study design and will be adjusted for in statistical analyses. For each centre patients will be allocated to one of the two treatment groups using a randomization list that was previously prepared by the study statistician. The list will be gerenated by blocked randomization. Sealed envelope will be used in each centre to ensure allocation concealment. Participant will be assigned for test or control treatment out between days -7/-10 and day 0. The therapist will be informed about treatment allocation by opening the envelope at the beginning of the treatment appointment.

Schedule for each visit

Participants who have expressed a degree of interest in participating from face-to-face discussions or from responses to advertisements will be invited to a Screening visit. This will take place, as all study visits will, at the Hospital General de Catalunya (Barcelona) and at the Odontostomatology Units (Clinica de Odontologia) of Madrid, Santiago de Compostela, Murcia and Granada, and this should take approximately 45 minutes. This will take place at a mutually convenient time and date for the potential participant and the study dentist, within the confines of clinical space availability. Here they will be initially asked about their personal information/medical history and undergo a dental examination. If they are eligible, they will be informed when the next stage of the study will commence and following an appointment is given in order to begin with the investigation. Treatment will be provided by the post-graduate students of the Master of Periodontology of each centre.

One-two weeks later on Day -7/-10 (baseline appointment or visit 1), informed consent will be given and signed. Blood, GCF, plaque and stool samples will be collected. Medical history, adverse events and concomitant medications will be checked and an oral examination will be carried out including recording number of teeth and at 6 sites per tooth probing depth, recession (mm) and bleeding after probing. A very superficial prophylaxis, motivation and oral hygiene instructions will be provided.

On Day 0 (morning) (visit 2), patients assigned to the test group will start the FMD for 5 consecutive days. All patients will undergo full-mouth subgingival instrumentation (PMPR) procedures and more detailed hygiene instruction will be reinforced. Medical history, adverse events and concomitant medications will be checked, and an oral examination will be carried out in order to screen for complications. A trained registered dietitian (from one of the centres) will discuss FMD with patients and also distribute survey to report items not eaten and extra food consumed.

On day 1 (v3), samples of blood and GCF will be taken. Medical history, adverse events and concomitant medications will be checked, an oral examination will be carried out in order to screen for complications.

On day 7 (v4), samples of blood and GCF will be taken. Medical history, adverse events and concomitant medications will be checked, an oral examination will be carried out in order to screen for complications.

On day 45±5 (v5), samples of blood and GCF will be taken. Oral hygiene instructions will be reinforced and a session of supragingival scaling with polishing will be provided. The second cycle of FMD will be started in patients of the test group. Medical history, adverse events and concomitant medications will be checked, an oral examination will be carried out in order to screen for complications.

On day 85 ±5 (v6), the third cycle of FMD will be started in patients of the test group. Medical history, adverse events and concomitant medications will be checked, oral hygiene instructions will be reinforced and a session of supragingival scaling with polishing will be provided.

On day 90 ±5 (v7), full-mouth periodontal charting measurements will be recorded. Samples of blood and GCF samples will be taken. Oral hygiene instructions will be reinforced and, if necessary, a session of supportive periodontal therapy will be provided. Medical history, adverse events and concomitant medications will be checked, an oral examination will be carried out in order to screen for complications.

On day 180 ±10 (v8), full-mouth periodontal charting measurements will be recorded at 6 sites per tooth: probing depth, recession (mm) and bleeding after probing. Blood, GCF, plaque and stool samples will be taken. Oral hygiene instructions will be reinforced. Medical history, adverse events and concomitant medications will be checked, an oral examination will be carried out in order to screen for complications.

*Patients will be called one or two times during each FMD cycle to check that everything is proceeding properly and to solve any problems or concerns they may have.

Follow up Procedures

If a participant misses multiple (2/3) visits they could be considered as a drop-out. However, they will be included in the intention-to treat analysis.

End of Study Definition

The study will be complete once all the participants have finished all the phases of the clinical period, and the processing/analysis on the biological material and clinical scores has been performed.

Sample Collection/Labelling/Logging

The samples will be collected during the study visit from the patient by qualified dentists of the International University of Catalunya, Complutense University of Madrid, University of Santiago de Compostela, University of Murcia and University of Granada who will participate in this study. During the collection of all sample types, proper hand hygiene, fitted gloves and sterile single-use examination items will be used to ensure the integrity of the samples collected and the safety of the examiner and participant. Pseudo-anonymised labelled tubes will be prepared in advance of each visit, with the label consisting of the participant number prefixed with the sample type designation e.g. G for GCF, B for blood, S for saliva, SubP for sub-gingival plaque etc. Collection of samples will take place at each visit before clinical examination takes place, to prevent the physical manipulation from disturbing the sampling site or from causing slight gingival bleeding which may contaminate the sample being collected. GCF Periopaper® Strips (Pro-flow Inc., Amityville, New York, USA) will be placed in the gingival crevice of the teeth with the deepest pocket site (buccal aspects) in each quadrant. They will then be immediately measured on a calibrated Periotron 8000 (Pro-Flow Inc., Amityville, New York, USA) electronic transducer, which will quantify the amount of GCF collected. Once measured, the GCF strips for that visit will all be stored at -80ºC in a single 2ml tube and pooled for further analysis. 4ml of venous blood will be collected from the participant's arm into Hemogard safety closure capped evacuated sterile vacutainers, containing the anticoagulant K2 Potassium salt of EDTA (Ethylene Diamine Tetra Acetic acid) that has been spray coated onto the interior surface of the tube. Samples will be taken by experienced and trained phlebotomists. To reduce this risk of fainting, participants will be on a semi- reclined plinth throughout the duration of the sampling and for five minutes following sampling. A researcher will be present with the participant at all times to ensure no falls or injuries are sustained in the event of fainting. Used needles will be discarded into a secure sharps bin. The samples for serum will be centrifuged for 10mins at 11,000 RPM then immediately divided into 0.2ml - 0.5ml aliquots and stored in a freezer at -80°C, until required for analysis. Sub-gingival plaque samples will be collected from the buccal surface of the tooth by the study dentist using a sterile curette, from below the gingival margin respectively. The plaque will be collected from teeth with the deepest pocket site (buccal surface) at each study visit. These teeth were selected to have a good mixture of molars and incisors. The collected plaque from these four teeth will be pooled into 1ml of sterile 0.1x Tris-EDTA and stored at -80ºC. Participants will be provided with home collection kits for sampling of stool in preserving solution ([http://www.microbiome-standards.org)] http://www.microbiome- standards.org) and this sample will be posted to the local laboratory within 7 days of collection. On receipt of stool samples in the laboratory, samples will be stored at -80 C. All biologically contaminated disposable items will be discarded into the correct biological hazard bin for processing and removal. All samples taken will be logged onto the participant's hardcopy CRF for that study visit, with the date and time of collection recorded and the initials of the collecting study dentist. This will also be logged onto the study Excel spreadsheet. If a particular sample is not able to be taken at that visit, the reason for this will be stated in the appropriate 'Additional notes' section of the CRF.

Sample Analysis Procedures

All experiments will be conducted in the Microbiome and Salivary laboratories, Guy's Hospital. GCF samples will be thawed and eluted in PBS (pH 7.2±0.2) supplemented with Easypack Protease Inhibitor Cocktail (Roche) as described in Curtis et al. 1988. Briefly, the periopaper strips will be placed in a perforated 0.5ml microcentrifuge tube which will be held inside a 1.5ml tube. The elution buffer (50μL) will be added on to the strips and placed in a vortex shaker for 2 minutes before centrifugation for 15 minutes at 11,000 rpm and 4 ̊C. The centrifugation will be repeated with a further 50μL of the elution buffer added on to the strips, to yield ~90μL of total eluted GCF. Protein concentration will be quantified using an LVis plate (BMG Labtech CLARIOstar) calibrated with Bovine Serum Albumin (Sigma). GCF analysis for selected analytes will be performed by Luminex. Samples will be processed at the KCL Centre for Host-Microbiome Interactions, fl.17 Guys Tower Wing. Plaque and stool samples will undergo DNA extraction following standard procedures in our lab and will be analyzed using next generation DNA sequencing to characterize the subgingival microbiota in order to identify and determine the levels of key periodontal bacterial pathogens and microbial community-wide changes in sites treated with both test and control protocols. Blood samples will be tested for cytokines, acute phase proteins and inflammatory markers using various techniques such as Western blots or enzyme-linked immunosorbent assays (ELISA), which will determine the presence and amount of these in the blood. Gingival Crevicular Fluid will be analysed for inflammatory mediators, antibodies, peptides and cytokines, again using techniques such as ELISA. Circulating levels of IGF-1, fasting blood glucose level, blood β-Hydroxybutyrate level will be assessed to monitor the compliance to FMD.

ELISA (high-sensitivity two-site enzyme-linked immunosorbent assay): IL-6 detection.

Cobas Integra 700 (automated immuno-turbidimetric high-sensitivity assay): HsCRP detection.

The data generated from these experiments will be stored on secure, password- protected King's computers, including those in the Salivary and Microbiome laboratories and the study laptop provided by King's.

Sample Storage Procedures

Blood, saliva, plaque and GCF samples will be stored at -80ºC in secure, locked HTA freezers in the laboratories of International University of Catalunya, Complutense University of Madrid, University of Santiago de Compostela and University of Granada. This will ensure long term stability in preparedness for sample processing. Following collection, stool samples will be sent to each participating centre by patients in sealed pre-stamped envelopes. As they are stored, all samples will have their physical integrity checked and samples to be frozen will then be logged onto a password-protected, secure computer database, which records their location in the freezer and the time/date they were stored. A physical hardcopy recording the samples being stored will also be featured on the CRF. The storage, transport, use and ultimate disposal of the sample provided will be conducted in compliance with the UK Human Tissue Act 2004 and with the EU Tissues and Cells Directives. If any samples are not immediately processed, they will be pseudo-anonymously stored for further analysis at a later date. Samples will be transferred to Salivary laboratory, Guy's Hospital and will be archived for 10 years after completion. After ethics approval for the study has expired, the blood, saliva and GCF samples will be disposed of in accordance with the Human Tissue Act 2004, and any amendments thereto, or transferred to a tissue bank.

Shipping of sample from Spain to UK

Samples will be placed in an igloo that can contains sufficient ice/dry ice to ensure samples are kept at the correct temperature for longer than the estimated journey time. Then, the polystyrene igloo is partially filled with ice/dry ice allowing room for samples and extra ice. Samples may be placed in a sealed plastic bag to aid cataloguing. The igloo is then filled with dry ice to cover the samples and a dispatch form and, additionally, a copy of the address label in a sealed plastic specimen bag is included. A lid will be placed on the igloo and secured with packing tape. Following that, the igloo is wrapped in strong brown wrapping paper and both an address label and very low temperature hazard labels are attached before the delivery. It will be selected the fastest mean of transport (e.g., plane) in order to complete the shipping as fast as possible.

Assessment of Safety

The investigators do not foresee any significant risks to the participant involved with the sample collection, including blood samples, as these are well-established procedures. Based on previous literature, a possible risk might concern some mild/moderate systemic adverse events caused by the FMD diet regimen, including fatigue, weakness and headaches. There is also a slight risk of fainting during or following blood sampling. To reduce this risk, participants will be on a semi-reclined plinth throughout the duration of the sampling and for five minutes following sampling. A researcher will be present with the participant at all times to ensure no falls or injuries are sustained in the event of fainting. If a needle stick injury occurs to the examiner during the collection of the blood sample, or a scratch injury occurs, local procedures will be implemented to respond to such an incident. No serious adverse events are expected to occur during the course of the study.

Ethics Reporting

An Adverse Event is any unfavourable and unintended signs, symptoms or disease associated with the study. Should an Adverse Event occur, such as fainting during the taking of blood, the investigator will inform the Chief Investigator, for inclusion in the study file CRF. A Serious Adverse Event (SAE) is an event that causes death, requires the hospitalisation of the participant, causes persistent disability, or causes a birth defect. Should this occur, a report will be logged within 24 hours of learning of the event and a report to the ethics committee within 15 days of learning of the event. The form should be completed in typescript and signed by the chief investigator. The main REC will acknowledge receipt of safety reports within 30 days.

Compliance and withdrawal

Subject compliance

Participant compliance will be assessed at each study visit. A self-reported medical history will ensure that the participant has not taken any action (e.g., started to participate in another clinical trial) or developed a condition or started taking medication (e.g. taking systemic antibiotics) which is prohibited by the exclusion criteria. This will be recorded on a checklist on the CRF. Each patient should fill a diet diary to throughout the study including FMD cycles for test patients. Failure to complete the dietary diary would also be recorded as drop-out, due to the crucial importance of diet for the validity of the study. Lastly, if a participant unexpectedly fails to attend a study visit, they will be requested to attend clinic at the very next possible opportunity.

Withdrawal / dropout of subjects

Participants may withdraw from the study at any time. This would be through a verbal discussion between the participant and any of the study team, and their decision logged on a written Withdrawal form. Reasons for withdrawal could be due to physical discomfort or too great a time commitment for example. Upon completion of the data analysis, where all anonymised data would be collated, participants would no longer be able to withdraw their data from the study, which would be made clear at the initial recruitment stage. The latest date for this is at the end of the study. Certain circumstances may require the study team to decide to withdraw participants from the trial, such as significant non-compliance to the protocol e.g., missing multiple study visits, or other events which would fulfil the exclusion criteria. This would involve speaking with the participant to inform and explain the decision to them, and the decision logged on a written Withdrawal form. If non-compliance is revealed at a study visit, it would also be logged in the 'Additional Notes' section of the CRF. Subjects will not be replaced when individuals withdraw.

Statistical considerations

Sample size calculation

No studies have been published using FMD in periodontitis patients. Therefore, no data about feasibility and required sample size is available in the literature. it is very difficult to estimate what the correct study sample size would be and, as a consequence, this study is designed as an internal pilot. While Browne and co-workers (1995) suggested 28 patients would be required as rule of thumb for sample size, Kieser & Wassmer (1996) found that a pilot sample size between 20 and 40 would minimise the overall sample size of the larger study. Following the suggestion by Julious 2009, 12 patients per study arm will be recruited for this study.

Interim analysis and feasibility/progression criteria

The decision to progress with the larger trial (and the relative sample size) will depend on the feasibility/progression criteria below.

FEASIBILITY ASPECTS PROGRESSION CRITERIA TO BE SATISFIED

Willingness to be randomized ≥ 50% of approached patients agree Self-reported compliance with diet ≥ 66% of test group patients self-report compliance (defined as not more than 1 day in which the diet was not followed)

Acceptance of blood samples ≥ 66% of recruited patients have all blood samples taken as per protocol Absence of serious adverse events No patients report serious adverse events which might be related to the test diet

If all criteria above are met, analysis of existing data up to 3 months will be carried out, using data from the 28 'internal pilot' patients. Means and standard deviations of hs-CRP values at 3-months will be used to calculate the required sample size for the larger trial. Follow-up of the study patients will continue up to 6 months post-treatment. Should the difference between groups for the primary outcome (hs-CRP at 3 months) be minimal, resulting in a very large sample size, a decision may be made not to progress to recruiting a larger group of patients and recruitment will be stopped. However, the patients still in the study will be followed up until the last study follow up (180 days).

Statistical analysis

The primary outcome of the study is circulating hs-CRP levels at 3 months post- treatment (test vs. control). However, the internal pilot/feasibility part of the study will need to completed first before considering whether to proceed with a fully-powered study sample size. If feasibility criteria are met, the difference in CRP levels at 3 months post-treatment between groups will be used to the sample size, and a formal statistical plan will be formulated. Different statistical packages will be used for different purposes, Stata 14 (StataCorp LLC, College Station, Texas, USA) will be main package and R (with R-Studio plugin), will be used for additional analyses, both of them with specific routines created for this study. The Shapiro-Wilk Test will be applied to verify if the quantitative variables analysed follow a normal distribution and logarithmic transformation will be performed in those that do not follow it. The profile of the population and of the study groups will be described. The results of the qualitative variables will be expressed in proportions and the quantitative variables will be expressed as means and standard deviation, including the 95% confidence intervals. The distribution of the population for each of the clinical, biochemical and microbiological parameters will also be obtained. For the bivariate analysis, chi-square test will be used to determine if there is a statistically significant association between two qualitative variables, the data will be presented as contingency tables, when the Chi- square test does not meet the validity conditions Fisher's exact test will be applied.

To compare the means of two independent variables for intergroup analyses, the Student's T-test will be used, considering Student's T-test for paired samples in within-group analyses. If the normal assumptions are not fulfilled, the No Parametric "Mann-Whitney U" test will be applied. For intragroups analyses, ANOVA for repetitive measures or Friedman test will be used. Multivariate analysis will be performed by means of a multiple linear regression model and ordinal logistic regression introducing in it the independent variables with a lower significance level of 0.20. The conditions will be checked by residual analysis of heteroscedasticity and linearity. The level of statistical significance for this study will be p<0.05.

Stopping / discontinuation rules and breaking of randomisation code

The investigators do not foresee any risks involved with the sample collection and FMD, as these are well-established procedures. Therefore, the investigators foresee no part of the study should need to be discontinued and the trial shouldn't need to be stopped due to participant safety concerns. However, since FMD has not been tested in periodontitis patients, in the unlikely event that there is a Serious Adverse Event, a report to the Sponsor will be logged within 24 hours of learning of the event and a report to the ethics committee within 15 days of learning of the event. A decision will then be made as to whether or not the study should stop in conjunction with these bodies.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years
* Periodontitis stages III-IV, generalized, grade C-B (according to the New World Workshop 2017)
* Minimum of 20 teeth present: to ensure there are sufficient teeth for study and that the same teeth can be examined in all participants.
* Systemically healthy participants (self-reported questionnaires will be used).
* Body mass index: 18.5-30 kg/m2 (normal weight to overweight, but not obese)
* Be willing and competent (verbally and cognitively) to give written informed consent and complete a medical history form
* Be willing and physically able to carry out all study procedures (e.g. multiple cycles of a 5-day dietary regimen and blood samples)
* Absence of hopeless teeth, acute dental conditions, teeth with endodontic-periodontal lesions and necrotising periodontal diseases

Exclusion Criteria:

* Age > 70 years. Exclusion for safety and feasibility reasons and to minimize the complicating factors such as frailty and un-/under-diagnosed medical conditions.
* Less than 20 teeth present
* Patients who received any periodontal treatment in the last 12 months
* Smoking (defined as self-reported use of any cigarettes or electronic cigarettes for at least 5 years): to avoid the potential confounding effect of smoking
* Mental illness, including severe depression, dementia. To ensure safety and compliance of the protocol
* Drug dependency
* Hormone replacement therapy (DHEA, estrogen, thyroid, testosterone).
* Severe hypertension (systolic BP > 200 mm Hg and/or diastolic BP > 105 mm Hg)
* Underweight (BMI < 18.5 kg/m2)
* Currently taking part in other clinical trials: to prevent either from interfering with the results of the other
* Pregnant or breastfeeding women: to prevent hormonal changes from influencing the amount of inflammation
* Taking medications including systemic anti-inflammatory medication within 3 months of the study (NSAIDs, no more than once per week and not in the week before sample collection, is permitted)
* Systemic antibiotic intake within 3 months: to prevent their microbiome-modulating effects from impacting the inflammatory status.
* Current orthodontic treatment: interferes with plaque control measures.
* Alcoholism (alcohol intake greater than two drinks per day for women and three drinks per day for men)
* Denture wearer/presence of dental implants: They may have an effect on periodontal parameters of neighbouring teeth
* Obvious signs of untreated caries and other significant oral diseases which in the opinion of the Study Dentist will affect either the scientific validity of the study, or if the volunteer was to participate in the study would affect their wellbeing
* Unable or unwilling to participate in baseline or follow-up examinations
* Unable or unwilling to complete the dietary intervention
* Special dietary requirements incompatible with the study interventions
* Significant food allergies which would make the subject unable to consume the food provided

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2023-12-04 (Actual); Primary Completion 2024-04-26 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
High-sensitivity C-reactive protein (hs-CRP) values in serum | It will be measured at baseline and 90 days after treatment.
  Blood samples will be taken. A multiple bead immunoassay technique (Luminex) will be used to detect the serum levels of CRP (as alternative ELISA technique may be used). CRP will be measured in milligrams of the protein per liter of plasma (mg/L).

SECONDARY OUTCOMES:
Hs-CRP values in serum | It will be measured at baseline and 1-, 7-, 45- and 180 days after treatment
  Blood samples will be taken. A multiple bead immunoassay technique (Luminex) will be used to detect the serum levels of CRP (as alternative ELISA technique may be used). CRP will be measured in milligrams of the protein per liter of plasma (mg/L).
Clinical attachment level (CAL) | It will be measured at baseline (before treatment) and 90- and 180 days after treatment
  CAL will be measured with a periodontal probe from University of North Carolina (UNC-15) and the values will be expressed in millimeters (mm).
Probing pocket depth (PPD) | It will be measured at baseline (before treatment) and 90- and 180 days after treatment
  PPD will be measured with a periodontal probe from University of North Carolina (UNC-15) and the values will be expressed in millimeters (mm).
Bleeding on probing (BOP) | It will be measured at baseline (before treatment) and 90- and 180 days after treatment
  BOP will be assessed dichotomously by assigning a binary score to each surface (1 for presence, 0 for absence)
Plaque index (PI) | It will be measured at baseline (before treatment) and 90- and 180 days after treatment
  PI will be assessed dichotomously by assigning a binary score to each surface (1 for presence, 0 for absence)
Inflammatory biomarkers from Gingival crevicular fluid (GCF) | GCF will be collected at baseline and 1-, 7-, 45- 90- and 180 days after treatment. Plaque and stool sample will be collected at Baseline and 180 days after treatment
  Luminex techniques for GCF will be used and biomarkers (Interleukin-1alfa (IL-1a),-1beta (IL-1b),-6 (IL-6),-10 (IL-10),-17 (IL-17), Leptin. Markers related to the response to FMD: Insulin like growth factor binding protein-1-to-6 (IGFBP-1-to-6) and Matrix metalloproteinase-8 (MMP-8) quantities will be expressed in ng/ml.
Sub-gingival plaque | Plaque will be collected at Baseline and 180 days after treatment
  DNA extraction protocols for plaque will be used to determine the presence of bacteria.
Stool samples | Stool sample will be collected at Baseline and 180 days after treatment
  DNA extraction protocols for stool will be used to determine the presence of bacteria
Patients reported outcome measurements (PROMs) | It will be measured at baseline, and 90- and 180- days after treatment
  An Oral Health-Related Quality of Life questionnaire with 14 items (OHIP-14) will be given to assess the quality of life related to people's perception of oral disorders on their well-being. In detail, responses will be coded 4="very often", 3 ="fairly often", 2 ="occasionally", 1="hardly ever" and 0="never". A lower score means a better outcome (e.g., 0 indicates that the patient has never experienced an unpleasant condition), whereas a higher score (e.g. 4) means the worst outcome

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Nibali, DDS, PhD, Principal Investigator — King's College London
Locations (5):
- Spain (5):
  - Universitat Internacional de Catalunya, Sant Cugat del Vallès, Barcelona
  - Universidad de Granada, Granada
  - Universidad Complutense de Madrid, Madrid
  - Universidad de Murcia, Murcia
  - Universida de Santiago de Compostela, Santiago de Compostela

IPD SHARING:
Plan to Share IPD: No
IPD will be not shared. Data will be anonymized. In the future publication data of each patient will be pooled with the ones of the other patients according to the statistics method that will be followed.

REFERENCES:
- [Background] Wei M, Brandhorst S, Shelehchi M, Mirzaei H, Cheng CW, Budniak J, Groshen S, Mack WJ, Guen E, Di Biase S, Cohen P, Morgan TE, Dorff T, Hong K, Michalsen A, Laviano A, Longo VD. Fasting-mimicking diet and markers/risk factors for aging, diabetes, cancer, and cardiovascular disease. Sci Transl Med. 2017 Feb 15;9(377):eaai8700. doi: 10.1126/scitranslmed.aai8700. PMID 28202779
- [Background] Longo VD, Di Tano M, Mattson MP, Guidi N. Intermittent and periodic fasting, longevity and disease. Nat Aging. 2021 Jan;1(1):47-59. doi: 10.1038/s43587-020-00013-3. Epub 2021 Jan 14. PMID 35310455
- [Background] Graziani F, Cei S, Tonetti M, Paolantonio M, Serio R, Sammartino G, Gabriele M, D'Aiuto F. Systemic inflammation following non-surgical and surgical periodontal therapy. J Clin Periodontol. 2010 Sep;37(9):848-54. doi: 10.1111/j.1600-051X.2010.01585.x. Epub 2010 Jun 4. PMID 20546085
- [Background] Machado V, Botelho J, Escalda C, Hussain SB, Luthra S, Mascarenhas P, Orlandi M, Mendes JJ, D'Aiuto F. Serum C-Reactive Protein and Periodontitis: A Systematic Review and Meta-Analysis. Front Immunol. 2021 Jul 28;12:706432. doi: 10.3389/fimmu.2021.706432. eCollection 2021. PMID 34394107
- [Background] Mainas G, Santamaria P, Ide M, Longo V, Vinciguerra M, Nart J, Nibali L. Could dietary restrictions affect periodontal disease? A systematic review. Clin Oral Investig. 2023 Aug;27(8):4107-4116. doi: 10.1007/s00784-023-05052-9. Epub 2023 May 18. PMID 37199773